CLINICAL TRIAL: NCT07198412
Title: Impact of Ultrasound-Guided Spinal Anesthesia and Pre-Procedure Sedation on Postoperative Acute and Chronic Back Pain in Non-Obstetric Surgery.
Brief Title: Effect of Sedation After Ultrasound-Guided Spinal Anesthesia on Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Samar Rafik Mohamed Amin, Assistant professor of anesthesia and intensive care, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RC_7.8.2025
Record Dates: First submitted 2025-09-15; First posted 2025-09-30 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Pain Management; Postoperative Acute Pain; Chronic Back Pain
Keywords: Spinal anesthesia; Ultrasound-guided anesthesia; Pre-procedure sedation; Midazolam; Chronic back pain
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A - Ultrasound-Guided Spinal Anesthesia (No Sedation) (Active Comparator)
  Interventions: Procedure: Ultrasound-guided spinal anesthesia
- Arm B - Ultrasound-Guided Spinal Anesthesia with Sedation (Midazolam) (Experimental)
  Interventions: Drug: Midazolam plus ultrasound-guided spinal anesthesia
- Arm C - Landmark-Guided Spinal Anesthesia (Control) (Placebo Comparator)
  Interventions: Procedure: Landmark-guided spinal anesthesia

INTERVENTIONS:
Procedure: Ultrasound-guided spinal anesthesia — Spinal anesthesia performed under real-time ultrasound guidance using a curvilinear ultrasound probe and 25-27G pencil-point spinal needle. Intrathecal injection of bupivacaine 0.5% hyperbaric (12-15 mg) following local infiltration with lidocaine 1% (2-3 mL).
  Arms: Arm A - Ultrasound-Guided Spinal Anesthesia (No Sedation)
Drug: Midazolam plus ultrasound-guided spinal anesthesia — Patients will receive midazolam (0.02-0.05 mg/kg IV; max 5 mg) 5-10 minutes prior to spinal anesthesia. Ultrasound guidance used for spinal needle placement. Intrathecal bupivacaine 0.5% hyperbaric (12-15 mg) after lidocaine 1% (2-3 mL) infiltration. Oxygen supplementation at 2 L/min and standard monitoring.
  Arms: Arm B - Ultrasound-Guided Spinal Anesthesia with Sedation (Midazolam)
Procedure: Landmark-guided spinal anesthesia — Spinal anesthesia performed using the traditional landmark palpation technique without ultrasound guidance or sedation. Intrathecal bupivacaine 0.5% hyperbaric (12-15 mg) after lidocaine 1% (2-3 mL) infiltration, using a 25-27G pencil-point spinal needle.
  Arms: Arm C - Landmark-Guided Spinal Anesthesia (Control)

SUMMARY:
This study will evaluate whether giving sedation before spinal anesthesia, when performed with ultrasound guidance, reduces the risk of developing back pain after surgery. Spinal anesthesia is commonly used but may cause discomfort or persistent back pain in some patients. By comparing standard techniques, ultrasound guidance, and sedation, we aim to find safer and more comfortable approaches for patients undergoing non-obstetric surgery.

DETAILED DESCRIPTION:
Spinal anesthesia is widely used for abdominal and lower limb surgeries, yet a significant number of patients experience new back pain afterward, sometimes lasting for months. Contributing factors include needle size, multiple puncture attempts, and patient characteristics. Ultrasound guidance can improve accuracy and reduce complications, while pre-procedure sedation may lower anxiety and discomfort during the procedure.

This randomized controlled trial will include 180 adult patients scheduled for non-obstetric surgery. Participants will be divided into three groups:

Ultrasound-guided spinal anesthesia without sedation

Ultrasound-guided spinal anesthesia with sedation (midazolam)

Landmark-guided spinal anesthesia (control)

Sedation will be administered with midazolam before the spinal procedure in the sedation group. All patients will receive standardized anesthesia techniques. Pain will be assessed in the early postoperative period and during long-term follow-up (1, 3, and 6 months) using validated pain scales and questionnaires. Secondary outcomes include pain severity, number of needle attempts, procedure time, patient satisfaction, and complications such as headache or nausea.

This study will clarify whether combining ultrasound guidance with pre-procedure sedation can reduce both acute and chronic back pain after spinal anesthesia, aiming to improve patient safety, comfort, and satisfaction.

ELIGIBILITY:
Inclusion Criteria

Adults aged 18-65 years ASA physical status I-II Body Mass Index (BMI) ≤ 35 kg/m² Scheduled for elective non-obstetric lower abdominal or lower limb surgery under spinal anesthesia Able to provide written informed consent

Exclusion Criteria

Contraindications to spinal anesthesia (e.g., coagulopathy, local infection at puncture site) Pre-existing chronic low back pain Chronic opioid use Known allergy or contraindication to study medications (bupivacaine, lidocaine, midazolam) Psychiatric or neurological disorders affecting pain perception or reporting Severe spinal deformities or history of previous spinal surgery Inability to comply with follow-up assessments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Back Pain | 24-48 hours postoperatively; 1 month, 3 months, and 6 months after surgery
  Presence of pain or discomfort at the lower back or puncture site, assessed using a pain body map and Numeric Rating Scale (0-10). Evaluations will be performed both in the early postoperative period and during follow-up.

SECONDARY OUTCOMES:
Severity of Postoperative Back Pain | 24-48 hours; 1 month, 3 months, and 6 months postoperatively
  Intensity of back pain rated using the Numeric Rating Scale (0-10).
Number of Needle Insertion Attempts | During the procedure
  Documented as single attempt versus multiple attempts (>2).
Patient Satisfaction | 24 hours postoperatively
  Patient-reported satisfaction assessed using a 5-point Likert scale.
Procedure-Related Complications | Within 7 days postoperatively
  Incidence of post-dural puncture headache, nausea, vomiting, urinary retention, or neurological deficits.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University Hospital, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No